CLINICAL TRIAL: NCT05047198
Title: Catheter Ablation Versus Radio-Ablation for Ventricular Tachycardia: a Randomized Controlled Trial
Acronym: CARA-VT RCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-2021
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Prospective, vanguard non-inferiority, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Catheter Ablation using invasive mapping
  Interventions: Procedure: Control - Catheter Ablation for VT
- Treatment (Experimental): Radio-ablation using non-invasive mapping
  Interventions: Procedure: Treatment - Non-Invasive Radio Ablation for VT

INTERVENTIONS:
Procedure: Control - Catheter Ablation for VT — Currently standard of care involves surgical resection of myocardial scarring in structural heart disease. Imaging is performed to identify culprit areas for ablation, pre procedural imaging involves echocardiography, CT scanning and PET imaging to assess cardiac function, ischemia, inflammation and scarring. Radiofrequency energy is delivered via catheter to the targets and is performed under sedation or anesthesia using multiple catheters placed in the heart while the patient is anticoagulated. A conventional approach will be used advancing multiple catheters via femoral veins and/or arteries under a combination of fluoroscopic, ultrasound and electroanatomic guidance. Ablation targets include an arrhythmogenic focus or the critical isthmus of the VT circuit and/ or substrate identified on preprocedural imaging or low voltage areas, "scar", identified during endocardial mapping. CA procedures for VT are often long, averaging approximately 5 hours .
  Arms: Control
Procedure: Treatment - Non-Invasive Radio Ablation for VT — Patients undergoing a non-invasive RA procedure for VT similarly require medical stabilization and multimodal imaging prior to treatment. A non-invasive electrophysiology study is performed under light sedation using ECGi mapping. This procedure requires only the placement of an IV cannula for light sedation, uses the ICD to stimulate VT which is mapped in real time using the ECGi mapping system. The multimodal imaging data is digitally fused and combined with the ECGi data to identify the VT circuit(s) and to attain the targets for radio-ablation. This analogue process is performed off-line by a physician team. The treatment plan is sent for alignment on a 4D planning CT performed with breath holding in the radiotherapy suite. Final treatment targets are reviewed by the local treating team and discussed with our collaborators remotely. Thereafter the patient is booked for a 15 minute out-patient radiotherapy treatment performed on a standard linear accelerator.
  Arms: Treatment

SUMMARY:
This study compares two arms - the current standard of care catheter ablation for Ventricular Tachycardia compared to stereotactic radiotherapy to non-invasively ablate ventricular tachycardia using a novel non-invasive ECG based body surface mapping technology. This allows investigators to identify ventricular tachycardia circuits to target for subsequent radio ablation. To summarize, the current standard of care invasive catheter ablation to the non-invasive radio ablation.

DETAILED DESCRIPTION:
Currently patients suffering Ventricular Tachycardia (VT) are offered drugs, such as Amiodarone, Implantable cardioverter defibrillatorf (ICD) implant and catheter ablation. Although effective drugs have side effects, ICD shocks are painful and catheter ablation is arduous for patients at high risk of complications. Catheter ablation is currently the gold standard treatment for recurrent VT despite anti-arrhythmic drugs (AADs).

Catheter ablation (CA) was initially developed in the 1980s following the successful treatment of VT by surgical resection of myocardial scarring in structural heart disease. After thorough clinical evaluation and medical stabilization, imaging is performed to identify culprit areas for ablation and to stratify risk of intervention. Pre procedural imaging in patients with ICDs in situ involves Echocardiography, Computerized Tomography (CT) scanning and Positron Emission Tomography (PET) imaging in order to assess cardiac function, ischemia, inflammation and scarring. If necessary mechanical circulatory support, Left Ventricular Assist Devices (LVAD) and/ or Extra Corporeal Membrane Oxygenation (ECMO) can be used to sustain cardiac output during VT induction and mapping.

Radiofrequency (RF) energy delivered via catheter to the arrhythmogenic target results in local resistive heating and is performed under sedation or anesthesia using multiple catheters placed in the heart while the patient is anticoagulated. Conventional approaches involve advancing multiple catheters via Femoral veins and/or arteries under a combination of fluoroscopic, ultrasound and electroanatomic guidance. Ablation targets include an arrhythmogenic focus or the critical isthmus of the VT circuit and/ or substrate identified on preprocedural imaging or low voltage areas, "scar", identified during endocardial mapping. CA procedures for VT are often long, averaging 5 hours duration reported in clinical trials, with prolonged procedures being associated with adverse outcomes and 30 day complication rates, including death, of 7- 13%.

Vulnerable patients requiring circulatory support or at high risk of recurrence and death following catheter ablation can be identified pre-operatively. Of all patients undergoing CA for VT, more than a third are "high risk" with a one year risk of death of >20%. Patients older than 65 with prior catheter ablation and recurrent VT with impaired left ventricular ejection fraction ≤35% have 90 day VT recurrence rates of 30% and mortality of 20%.

Patients with comorbidities such as Diabetes or COPD and those presenting in VT storm are also at high risk of hemodynamic compromise and death following Catheter Ablation. Without prophylactic LVAD placement, patients at high risk of haemodynamic instability (PAINESD score ≥ 15) suffer 30% death at thirty days with 41% VT recurrence post CA. It is these "high risk" patients that we believe will benefit from a non-invasive RA approach.

Patients undergoing a non-invasive Radio-Ablation (RA) procedure for VT similarly require medical stabilization and multimodal imaging prior to treatment. Instead of an invasive catheter-based electrophysiology study (EPS) and ablation, a non-invasive EPS (NIPS) is performed under light sedation using ECGi mapping. This short procedure, averaging 40 minutes, requiring only the placement of an IV cannula for light sedation, uses the ICD to stimulate VT which is mapped in real time using the CardioInsight ECGi mapping system.

The multimodal imaging data is digitally fused and then combined with the ECGi data to identify the VT circuit(s) and to target the arrhythmogenic tissue for radio-ablation. This analogue process is performed off- line by a committee of Cardiac Imaging and EP Cardiologists and a Radiation Oncologist. Once the target(s) are identified, the treatment plan is sent to Medical Physics for alignment on a 4D planning CT performed with breath holding in the radiotherapy suite. Final treatment targets are reviewed by the local treating team and discussed with our collaborators in St Louis. Thereafter the patient is booked for a 15 minute out-patient radiotherapy treatment performed on a standard linear accelerator.

Photon radiotherapy, as commonly used in cancer therapeutics across Canada, is guided using a cone beam onto the cardiac target(s). A single fraction of 25 Gy is delivered painlessly over 15 minutes. Although minor side effects have been reported, serious adverse events are rare and no ICD related issues have been described. No deleterious effects on cardiac function (LVEF) have been observed although approximately (5/65? TBC) patients have required a two week course of oral glucocorticoid therapy for symptomatic inflammation such as pericarditis or pneumonitis post RA25. All patients are treated with Rivaroxaban 20 mg po as prophylaxis against thromboembolism for thirty days post RA.

Radioablation is a novel procedure and long-term outcomes remain unknown. Reduction in VT is reported to be 85-92% up to 6 months post RA and in the ENCORE -VT study 17 of 19 patients were free from ICD shocks at 6 months. In the only prospective study of RA for VT, patients reported an improvement in quality of life in 5 of 9 domains remaining unchanged in 4. Long term safety data continue to be collected but cardiac irradiation <40 Gy has been historically associated with an approximate 1% excess mortality over years to decades in those receiving treatment for breast or lung cancer. This is in the context of a total mortality of 28% over 24 months of follow up in those undergoing CA for recurrent VT in Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥55 years of age
2. Cardiomyopathy (Left ventricular ejection fraction ≤ 35% and ICD in situ) AND
3. Recurrent VT events despite previous CA OR
4. VT events requiring intervention and PAINESD score ≥ 15

Exclusion Criteria:

1. Patients with NYHA Class IV heart failure &/ or with LVAD in situ
2. Patients not expected to live for more than one year for any reason
3. Patients who have previously received thoracic radiotherapy
4. Patients who are enrolled in another randomized clinical trial
5. Patients who are unable or unwilling to provide informed consent
6. Patients aged ≤54 years of age
7. Pregnancy (all women of child bearing age and potential will have a negative β-HCG test before enrollment)
8. Breastfeeding
9. Women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception (IUD, sterilization, birth control implant or birth control pill) throughout the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to composite event | 14 days
  Composite event including death at any time, appropriate ICD shock after 14 days, ventricular tachycardia storm after 14 days, treated sustained ventricular tachycardia below the detection rate of the ICD after 14 days

SECONDARY OUTCOMES:
Appropriate ICD ATP at any time or after 14 days | at any time or after 14 days
  Any appropriate therapy delivered from the ICD at least 14 days post randomization
Appropriate shocks | at any time or after 14 days
  Appropriate ICD shocks at any time post randomization
VT storm at any time or after 14 days | at any time or after 14 days
  3 or more episodes of VT occurring within 24 hours at any time post randomization
Sustained VT not treated by ICD at any time or after 14 days | at any time or after 14 days
  Time to sustained VT treated with appropriate any type of manual cardioversion after 14 days Any sustained VT greater than 30 seconds requiring manual cardioversion (ICD, external or pharmacologic)
Inappropriate ICD shocks at any time or after 14 days | at any time or after 14 days
  All inappropriate shocks from the ICD at any time post randomization
Any ICD shock at any time or after 14 days | at any time or after 14 days
  Both appropriate and inappropriate shocks from the ICD at any time post randomization
Any ventricular arrhythmia event at any time or after 14 days | at any time or after 14 days
  All ventricular arrhythmias including a composite of: appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion), VT storm/incessant VT.
  (composite of appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion)
Number of ICD shocks (all cause) | 3 years
  The number of all shocks from any cause will be calculated
Number of Anti-tachycardia pacing (ATP) | 3 years
  The total of all ATP delivered from the ICD will be calculated
Number of ICD appropriate therapy | 3 years
  Total number of therapies which received appropriate ICD therapy
Number of VT storm events | 3 years
  Total number of VT storms (3 episodes of VT within 24 hours)/ incessant VT will be calculated
Number of ventricular arrhythmia events | 3 years
  This is a composite of appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion, or VT storm/incessant VT. VT events which do not terminate despite exhausting ICD therapies will be considered incessant VT and included within the definition of VT storm.
Hospital admission for cardiac causes | 3 years
  Hospitalizations greater than 24 hours due to a cardiovascular cause.
Heart Failure decompensation /death | 3 years
  LVEF and RVEF assessed on 6-month and 24 month echocardiogram (absolute and delta compared to baseline).
Procedural complications and/ or antiarrhythmic drug adverse effects | 3 years
  and Periprocedural complications and adverse drug reactions will be assessed, any dose change or discontinuation of anti-arrhythmic medication due to abnormal blood tests (including kidney function, liver function, thyroid function) or any perceived side effects.
Patient Quality of life - SF36 | 3 years
  Will include responses from the Short Form 36
Cost-effectiveness | 3 years
  Quality adjusted life years (QALYs) will be derived from the case report forms and the questionnaires
Escalation and De-escalation of antiarrhythmic medication | 3 years
  Any increase or decrease in the dosage of antiarrhythmic medication either due to inefficacy or side effects will be assessed and reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Calum Redpath, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No